CLINICAL TRIAL: NCT01411644
Title: Phenotyping and Genotyping of Women Presenting With Ovarian Dysfunction Associated With a Hypergonadotropic Hypo-estrogenic Hormonal Status (WHO III) and Their First and Second Degree Relatives
Brief Title: Pheno- & Genotyping POF (WHO III)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Erasmus Medical Center (Other); Medical Center Alkmaar (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Medisch Spectrum Twente (Other); Isala (Other); Department of Clinical Pharmacy, University Medical Centre St Radboud, The Netherlands. (Other); Amphia Hospital (Other); Deventer Ziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Academisch Ziekenhuis Maastricht (Other); Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, professor, UMC Utrecht
Other Study IDs: METC 05-047
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Premature Ovarian Failure (POF); Incipient Ovarian Failure; Poor Response After Ovarian Hyperstimulation; Early Menopause; Hypergonadotropic Amenorrhea
Keywords: POF; IOF; Poor response; early menopause; Primary amenorrhea
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum and litium heparine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study focuses on the phenotyping and genotyping of women with hypergonadotropic ovarian dysfunction (WHO III status).

DETAILED DESCRIPTION:
First goal of the study is to phenotype patiens with hypergonadotropic ovarian dysfunction (WHO III) adequately. This group includes women with premature ovarian failure (POF), incipient ovarian failure (IOF), poor response after ovarian hyperstimulation, early menopause and hypergonadotropic primary amenorrhea. The standardized phenotyping consists of a questionnaire focusing on reproductive, medical, and family history; ultrasonography to assess ovarian reserve and/or antral follicle count and obtaining an extra blood sampling during routine endocrine screening for genotyping.

Phenotyping of patients presenting with ovarian dysfunction is of crucial importance when genotyping will be performed. The goal of this genotyping will be the identification of genetic factors associated with the (premature) depletion of the stock of ovarian follicles. It will be performed for isolated WHO III patients in an association (case-control) study for known candidate genes. In familial WHO III cases, genome wide linkage analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* POF; defined as secondary amenorrhea before 40 years of age and basal FSH > 40 IU/L
* Incipient ovarian failure; defined as normo-ovulatory cycles, raised basal FSH > 12 IU/L
* Poor response patients; defined as less than 4 oocytes retrieved or cancellation in case of absent follicle growth after ovarian hyperstimulation with 300 IU gonadotropins or cancellation in case of absent follicle growth
* Women with early menopause (between 40-45 years)
* Hypergonadotropic primary amenorrhea

Exclusion Criteria:

* Primary amenorrhea with early development disorders causing absence of ovaries and Swyer syndrome (XY)

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with WHO III status who attend the outpatient clinic of participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2005-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bart CJ Fauser, MD PhD, Study Director — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Knauff EA, Franke L, van Es MA, van den Berg LH, van der Schouw YT, Laven JS, Lambalk CB, Hoek A, Goverde AJ, Christin-Maitre S, Hsueh AJ, Wijmenga C, Fauser BC; Dutch POF Consortium. Genome-wide association study in premature ovarian failure patients suggests ADAMTS19 as a possible candidate gene. Hum Reprod. 2009 Sep;24(9):2372-8. doi: 10.1093/humrep/dep197. Epub 2009 Jun 9. PMID 19508998
- [Result] Knauff EA, Westerveld HE, Goverde AJ, Eijkemans MJ, Valkenburg O, van Santbrink EJ, Fauser BC, van der Schouw YT. Lipid profile of women with premature ovarian failure. Menopause. 2008 Sep-Oct;15(5):919-23. doi: 10.1097/gme.0b013e31816b4509. PMID 18551082
- [Result] Knauff EA, Eijkemans MJ, Lambalk CB, ten Kate-Booij MJ, Hoek A, Beerendonk CC, Laven JS, Goverde AJ, Broekmans FJ, Themmen AP, de Jong FH, Fauser BC; Dutch Premature Ovarian Failure Consortium. Anti-Mullerian hormone, inhibin B, and antral follicle count in young women with ovarian failure. J Clin Endocrinol Metab. 2009 Mar;94(3):786-92. doi: 10.1210/jc.2008-1818. Epub 2008 Dec 9. PMID 19066296
- [Result] Janse F, Knauff EA, Niermeijer MF, Eijkemans MJ, Laven JS, Lambalk CB, Fauser BC, Goverde AJ; Dutch Premature Ovarian Failure Consortium. Similar phenotype characteristics comparing familial and sporadic premature ovarian failure. Menopause. 2010 Jul;17(4):758-65. doi: 10.1097/gme.0b013e3181cf8521. PMID 20395876
- [Result] Knauff EA, Blauw HM, Pearson PL, Kok K, Wijmenga C, Veldink JH, van den Berg LH, Bouchard P, Fauser BC, Franke L; Dutch Primary Ovarian Insufficiency Consortium. Copy number variants on the X chromosome in women with primary ovarian insufficiency. Fertil Steril. 2011 Apr;95(5):1584-8.e1. doi: 10.1016/j.fertnstert.2011.01.018. Epub 2011 Feb 12. PMID 21316664